CLINICAL TRIAL: NCT00912613
Title: ICU Diaries as a Therapeutic Intervention for Post Traumatic Stress Disorder Following Critical Illness
Brief Title: Intensive Care Unit (ICU) Diaries as a Therapeutic Intervention for Post Traumatic Stress Disorder (PTSD) Following Critical Illness
Acronym: RACHEL II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: St Helens & Knowsley Teaching Hospitals NHS Trust (Other); Vrinnevishuset, Sweden (Unknown); Università degli Studi di Ferrara (Other); University of Copenhagen (Other); Haukeland University Hospital (Other); Hospital Pedro Hispano (Other); Sahlgrenska University Hospital (Other); General Hospital of Santo António (Other)
Responsible Party: Professor Richard David Griffiths, School of Clinical Science, University of Liverpool, Liverpool, UK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06/Q1502/127
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Critical illness; ICU Diaries; Post Traumatic Stress Disorder; Incidence
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Discussion with nurse (No Intervention): Brief discussion with ICU follow-up nurse about the patients' critical illness
- ICU Diary (Experimental): Receipt of ICU Diary at 1 month post critical illness
  Interventions: Other: ICU Diary

INTERVENTIONS:
Other: ICU Diary — ICU Diary containing daily information of patients condition and treatment with appropriate photographs
  Arms: ICU Diary

SUMMARY:
The incidence of PTSD post ICU varies from unit to unit, however a significant number of patients have been shown to develop this disorder. Many patients do not recall their stay in ICU properly and yet can clearly recall nightmares, hallucinations or paranoid delusions, which may be very frightening for the patient to recall at a later stage. As yet, no interventional studies have had an impact on the development of PTSD in this population of patients. However, a recent observational multi-centre study suggested that those patients receiving a diary of their time in ICU had lower levels of symptoms of PTSD than those who did not. These results need to be verified in the form of a randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Patients staying on the ICU for at least 72 hours (with greater than 24 hours of artificial ventilation)

Exclusion Criteria:

* ICU stay < 72 hours
* Too confused for informed consent
* Pre-existing psychotic illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Diagnosis of Post Traumatic Stress Disorder | 3 months post critical illness

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Griffiths, MD, Principal Investigator — University of Liverpool

REFERENCES:
- [Derived] Jones C, Backman C, Capuzzo M, Egerod I, Flaatten H, Granja C, Rylander C, Griffiths RD; RACHEL group. Intensive care diaries reduce new onset post traumatic stress disorder following critical illness: a randomised, controlled trial. Crit Care. 2010;14(5):R168. doi: 10.1186/cc9260. Epub 2010 Sep 15. PMID 20843344